CLINICAL TRIAL: NCT05590988
Title: Sensorimotor Arm Rehabilitation After Stroke Using Tablet-based Bimanual Coordination Training
Brief Title: Sensorimotor Arm Rehabilitation After Stroke
Acronym: TAB-APP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BDH-Klinik Hessisch Oldendorf (Other)
Collaborators: Gottfried Wilhelm Leibniz Universität Hannover (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TAB-APP
Record Dates: First submitted 2022-10-13; First posted 2022-10-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Hemiparesis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Results are evaluated by an independent scientists and group assignment is pseudonymised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tablet (Experimental): The intervention group trained bimanual coordination once a day for about 31 minutes on a total of ten days using a tablet game. A ball is to be moved on a circular line.
  Interventions: Other: Tablet-based training
- Aximo (Active Comparator): The patients in the control group receive an ergotherapeutic therapy unit once a day for the same length of time (approx. 31 minutes) for a total of ten days, in which they train unilaterally. In this therapy unit, the control group uses the "Aximo". This is a comb stand and so-called "rolls" with which plugging tasks can be practiced. The patients should push the rolls into the stand fields with the affected hand. With the plug-in game, the patients can complete different tasks that challenge and train their hand-eye coordination, their fine motor skills and their ability to grasp things (e.g. following a specific pattern based on a template or putting colors in a specific order).
  Interventions: Other: ergotherapeutic training

INTERVENTIONS:
Other: Tablet-based training — Each task is performed for one minute, followed by a 2-minute break. After the task has been performed three times, there is a 5-minute break. The training block is then carried out twice more. This means that three "blocks" are carried out for each therapy unit.
  Arms: Tablet
Other: ergotherapeutic training — A task is performed for one minute at a time, followed by a 2-minute break. Once three rounds have been completed, there is a 5-minute break. As in the intervention group, there are a total of three training blocks.
  Arms: Aximo

SUMMARY:
Hemiparesis is a frequently observed symptom of stroke. There are various therapy options that are used in the rehabilitation of patients. Some studies have shown that, in addition to unilateral arm training, bilateral arm training can also lead to positive results in treatment and is a useful addition to therapy. The newly developed app requires the coordination of both arms in certain time sequences and intensities or rhythms and addresses different sensory modalities (visual, auditory and kinesthetic). The aim of the study is to examine whether tablet-based training improves bimanual coordination.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an ischemic/hemorrhagic stroke
* moderate upper extremity paresis: 30 to 60 cubes in the Box-and-Block Test (BBT)
* sufficient resilience / alertness (active participation possible for at least 30 minutes)
* ability to give consent (written declaration of consent from the patient)

Exclusion Criteria:

* Hemianopia and/or neglect
* duration of illness >3 months
* pre-existing hemiparesis
* participation in another clinical trial within the last 30 days
* a pregnancy or breast-feeding period
* contraindications for MRI: claustrophobia; metallic or magnetic implants that contain iron, cobalt or nickel (e.g. pacemakers, brain pacemakers, automatic insulin pumps, electrodes, plates, clips, implanted hearing aids, dental implants, metal endoprostheses, metal parts or metal splinters in the body)

Ages: 36 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change of the hand/arm motor skills (unilateral) | Pre-test (day 1), Post-test (day 18), Follow-Up (day 25)
  measured by the difference in moving wooden cubes in the Box-and-Block Test (BBT) The BBT measures unilateral gross manual dexterity. The patient has to move as many individual cubes as possible from one side of the box over a partition to the other within one minute. The test takes place in a seated position and is performed sequentially with the non-impaired hand and the affected hand. The number of cubes transported for each side is evaluated.
Changes in bimanual coordination 1 | Pre-test (day 1), Post-test (day 18), Follow-Up (day 25)
  measured by the difference in moving wooden cubes in the modified Box-and-Block Test (mBBT) For this, a modified box with three compartments and two partitions is used. The task is to take a cube in one hand, pass it to the other hand over the first partition and then transport it over the second partition to the outer compartment. The dice are then counted in the outer compartment. The dice that fall from one hand to the other in the middle compartment are counted separately. The task is performed twice, starting with the unimpaired hand in the first run and with the impaired hand in the second run. The subject has one minute per round to transport as many cubes as possible to the outer compartment.
Changes in bimanual coordination 2 | Pre-test (day 1), Post-test (day 18), Follow-Up (day 25)
  measured by the difference in activity index (calculated from acceleration, movement amplitude and movement frequency during the use of the tablet game)

SECONDARY OUTCOMES:
Change of functional abilities | Pre-test (day 1), Post-test (day 18), Follow-Up (day 25)
  measured by the difference of National Institutes of Health Stroke Scale (NIHSS)
Change of activities of daily living | Pre-test (day 1), Post-test (day 18), Follow-Up (day 25)
  measured by the difference of Barthel-Index (BI)
Change of hand strength | Pre-test (day 1), Post-test (day 18), Follow-Up (day 25)
  Hand strength is measured with a KERN MAP digital hand force gauge. The change of strength (in kg) is calculated.
Change of selective motor control after a stroke | Pre-test (day 1), Post-test (day 18), Follow-Up (day 25)
  measured by the difference of the values of the "Fugl-Meyer-Test" (FMT)

OTHER OUTCOMES:
Change of functional connectivity of the motor system | Pre-test (day 1), Post-test (day 18)
  measured by differences between resting state functional magnetic resonance imaging (fMRI) scans

CONTACTS AND LOCATIONS:
Overall Officials: Jens D Rollnik, Prof. Dr., Principal Investigator — BDH-Klinik Hessich Oldendorf
Locations (1):
- Institute for Neurorehabilitation Research, BDH-Clinic Hessich Oldendorf, Hessisch Oldendorf, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No